CLINICAL TRIAL: NCT06748859
Title: The Effect of Iliopsoas Strain-counterstrain Technique on Mechanical Chronic Low Back Pain and Lumbar Flexion Restriction
Brief Title: Iliopsoas Counterstrain and Mechanical Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Javad Hassanzadeh, MSc. candidate of physiotherapy, Marmara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024/44-53
Record Dates: First submitted 2024-12-13; First posted 2024-12-27 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Mechanical Low Back Pain; Chronic Low Back Pain (CLBP)
Keywords: Mechanical chronic Low Back Pain; Myofascial Pain Syndromes; Strain-counterstrain; Psoas Muscles
MeSH Terms: conditions — Low Back Pain; Myofascial Pain Syndromes | interventions — Exercise Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Strain-counterstrain technique (Experimental): Participants in this group will receive strain-counterstrain technique and exercise therapy within two weeks.
  Interventions: Other: Counterstrain technique
- Exercise therapy (Active Comparator): Participants in this group will receive exercise therapy within two weeks.
  Interventions: Other: Exercise therapy

INTERVENTIONS:
Other: Counterstrain technique — In this group, participants will receive counterstrain technique on the Psoas major muscle and exercise training within two weeks.
  Arms: Strain-counterstrain technique
Other: Exercise therapy — participants who will assign to this group will receive exercise therapy within two weeks.
  Arms: Exercise therapy

SUMMARY:
The aim of this study is to determine the effects of the Strain-Counterstrain (SCS) technique on alleviating sudden and mechanical chronic low back pain and resolving limited lumbar flexion and extension in individuals with mechanical chronic low back pain (MCLBP), focusing on tender points in the Iliopsoas muscle. Our study is a randomized controlled trial. Based on sample size calculation, 32 voluntary patients with chronic mechanical low back pain will be recruited to the study. They will be then randomized into two groups using the Block Balanced Randomization method.

In the control group, consisting of 16 participants, 4 general exercises aimed at relieving back pain will be performed under the physical therapist's supervision. In the treatment group, also comprising 16 participants, after performing the exercises applied to the control group, the SCS technique will be applied to the tender points in the iliopsoas muscle: 90 seconds in a position of comfort, with 30-second intervals, 3 times on the more tender side and 2 times on the less tender side.

The assessment of the cases will use the visual analog scale (VAS) for pain intensity at rest and during lumbar flexion movement as primary outcome measurements TiltMeter© Application for joint range of motion (ROM), Modified Schober's Test (MST) for spinal mobility, Thomas test for iliopsoas muscle length, the Oswestry Disability Index (ODI) for stability, and 36-Item Short Form Survey (SF-36) for health-related quality of life. Assessments will be conducted before treatment, at the end of the 1st session, and at the end of the treatment (after six sessions). Significant results may reduce the burden on the healthcare system with the ease of application and low-cost advantage of the SCS technique, making treatment processes more efficient.

DETAILED DESCRIPTION:
Low back pain is one of the leading causes of disability and has been shown to occur more frequently than other health problems. When low back pain becomes chronic, the pain may often be less intense. Chronic low back pain is defined as pain that persists for more than 12 weeks. Many professionals and individuals working in demanding jobs often experience Chronic Non-Specific Low Back Pain, which results in reduced work capacity and significant impairment in daily activities. Additionally, many patients report increased pain while sitting or transitioning from a seated to a standing position.

Despite the rising number of patients presenting to hospitals with low back pain, the exact underlying cause is often not well understood. Recent studies suggest that most cases are due to mechanical causes, potentially resulting from improper biomechanical alignment.

The spinal curves, known as lordosis and kyphosis, play a critical role in energy expenditure and mobility from a biomechanical perspective. Improper adaptations and tensions between muscles can lead to either a loss or increase in lumbar lordosis, which can alter biomechanical structure and affect muscle function and range of motion. The psoas major muscle, which attaches to the L1-L5 vertebrae, can also influence lumbar lordosis if it becomes shortened.

Low back pain is typically nonspecific or mechanical. Mechanical chronic low back pain (CLBP) arises from the spine, intervertebral discs, or surrounding soft tissues due to excessive strain or injury. The iliopsoas muscles, deep muscles rarely stretched during daily activities, can become tense and contribute to this pain. As one of the strongest hip flexors, the iliopsoas plays a significant role in pelvic movement and stabilization. Tightness in the iliopsoas is often closely linked to low back pain. A shortened iliopsoas group may result in hyperlordosis, anterior pelvic tilt, and increased pressure on the spinal muscles. If the iliopsoas muscles are excessively tight, they can pull and twist the vertebrae, leading to disc compression and dysfunction, which may manifest as low back pain and discomfort around the sacroiliac joint. Research has found that individuals who work at desks often have shortened iliopsoas muscles, which can predispose them to future low back pain.

Individuals who sit for extended periods, such as sedentary workers and students, are at increased risk of musculoskeletal problems and muscle shortening. Research has shown that sitting for more than eight consecutive hours can lead to low back pain. The iliopsoas muscle, due to its unique connection between the lumbar spine and hip joint, is an important hip flexor affected by prolonged sitting. Biomechanical and electromyography studies suggest that control of the spinal curve is primarily provided by the psoas major muscle. When other muscles become less active, the psoas major becomes more engaged, helping to maintain an upright spine; however, a shortened psoas can lead to pelvic tilt and back pain.

Given the above reasons, many studies have been conducted to address iliopsoas muscle tightness. Research comparing techniques such as Proprioceptive Neuromuscular Facilitation (PNF) and Muscle Energy Technique (MET) for stretching the iliopsoas found that PNF was more effective, emphasizing the benefits of active mobilization and autonomic inhibition. However, muscle tightness can also originate from tender points, which, when addressed, can enhance proprioceptive activity and reduce hypersensitivity once the joint returns to its normal position. Despite the biomechanical importance of the iliopsoas muscle, research specifically focusing on tender points in this muscle remains limited.

Strain-Counterstrain is an osteopathic manipulation technique and the fourth most commonly used soft tissue method after High Velocity Low Amplitude (HVLA) and Muscle Energy Techniques (MET). This technique involves passive positional mobilization designed to alleviate musculoskeletal pain. Strain-Counterstrain helps correct neuromuscular imbalances caused by prolonged muscle stimulation. It is based on the proprioceptive theory, which suggests that this technique can rectify abnormal neuromuscular activity, often caused by sympathetic nervous system responses or inflammatory reactions. Studies have shown that the Strain-Counterstrain technique effectively restores range of motion and reduces pain in the lumbar region. Additionally, it is a low-cost, non-invasive treatment method. For example, a study demonstrated that both SCS and MET were effective in reducing pain and improving functional capacity in patients with chronic low back pain. Other research has reported positive effects on lumbar range of motion, pain, and quality of life when SCS was combined with techniques such as MET or McKenzie.

Most studies have focused on the quadratus lumborum muscle or general SCS techniques, and although the iliopsoas muscle is critically important, it has been less frequently studied in conjunction with SCS. Our study aims to clearly demonstrate the immediate and long-term effects of the iliopsoas-specific SCS technique on lumbar range of motion and pain, ultimately reducing the burden on healthcare systems in terms of labor and cost.

Hypotheses:

Null Hypothesis (H0): The Strain-Counterstrain technique has no positive effect on pain and restricted lumbar flexion in patients with chronic low back pain and limited lumbar flexion.

Alternative Hypothesis (H1): The Strain-Counterstrain technique has a positive effect on pain and restricted lumbar flexion in patients with chronic low back pain and limited lumbar flexion.

ELIGIBILITY:
Inclusion criteria:

1. Patients with chronic mechanical low back pain (CMLBP) aged between 18-60 years old;
2. Pain experience more than 12 weeks;
3. Pain intensity ≥ 3 based on Numeric pain scale;
4. Pain experience during lumbar flexion movement;
5. Positive Thomas test;
6. Having tenderness on Psoas major muscle 4 times more than palpation on ipsilateral quadratus lumborum muscle;
7. Able to understand and make communication with research team without any barrier;
8. Having consent to participate the study.

Non-inclusion criteria:

1. Pregnancy;
2. Not indicated for lumbar surgery based on diagnosis of a physical medicine and rehabilitation specialist,
3. Any type of fracture or history of trauma which makes manual therapy contraindicated for the patient,

Exclusion criteria:

1. Willing to discontinue the study progress for any reason;
2. Progressive deterioration during the study and intervention application.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2024-12-25 (Actual); Primary Completion 2025-02-23 (Actual); Study Completion 2025-03-05 (Actual)

PRIMARY OUTCOMES:
visual analog scale at rest | Baseline
  It is a commonly used tool for measuring pain. The patient is asked to mark their pain level on a 100-mm line, and the marked distance is then measured with a ruler from the left end and recorded. The scale typically ranges from zero, indicating no pain, to the highest, representing the most severe pain.
visual analog scale at rest | 30 minutes
  It is a commonly used tool for measuring pain. The patient is asked to mark their pain level on a 100-mm line, and the marked distance is then measured with a ruler from the left end and recorded. The scale typically ranges from zero, indicating no pain, to the highest, representing the most severe pain.
visual analog scale at rest | 2 weeks
  It is a commonly used tool for measuring pain. The patient is asked to mark their pain level on a 100-mm line, and the marked distance is then measured with a ruler from the left end and recorded. The scale typically ranges from zero, indicating no pain, to the highest, representing the most severe pain.
visual analog scale during lumbar flexion | Baseline
  It is a commonly used tool for measuring pain. The patient is asked to mark their pain level on a 100-mm line, and the marked distance is then measured with a ruler from the left end and recorded. The scale typically ranges from zero, indicating no pain, to the highest, representing the most severe pain.
visual analog scale during lumbar flexion | 30 minutes
  It is a commonly used tool for measuring pain. The patient is asked to mark their pain level on a 100-mm line, and the marked distance is then measured with a ruler from the left end and recorded. The scale typically ranges from zero, indicating no pain, to the highest, representing the most severe pain.
visual analog scale during lumbar flexion | 2 weeks
  It is a commonly used tool for measuring pain. The patient is asked to mark their pain level on a 100-mm line, and the marked distance is then measured with a ruler from the left end and recorded. The scale typically ranges from zero, indicating no pain, to the highest, representing the most severe pain.

SECONDARY OUTCOMES:
thomas test | Baseline
  The Thomas test is a method used to evaluate the shortening of the Iliopsoas muscle. There is no shortening if the tested leg is completely parallel to the bed. However, if the leg remains elevated from the bed, the angle should be recorded with a goniometer.
thomas test | 30 minutes
  The Thomas test is a method used to evaluate the shortening of the Iliopsoas muscle. There is no shortening if the tested leg is completely parallel to the bed. However, if the leg remains elevated from the bed, the angle should be recorded with a goniometer.
thomas test | 2 weeks
  The Thomas test is a method used to evaluate the shortening of the Iliopsoas muscle. There is no shortening if the tested leg is completely parallel to the bed. However, if the leg remains elevated from the bed, the angle should be recorded with a goniometer.
Modified Schober's Test | Baseline
  It is a commonly used method for assessing lumbar mobility. The patient stands with their feet shoulder-width apart, and a mark is placed between two posterior superior iliac spines (PSIS), adding 15 cm to it. The patient is then instructed to bend forward without bending their knees. The new distance between the two points is measured again, 15 cm is subtracted, and the result is recorded.
Modified Schober's Test | 30 minutes
  It is a commonly used method for assessing lumbar mobility. The patient stands with their feet shoulder-width apart, and a mark is placed between two PSIS, adding 15 cm to it. The patient is then instructed to bend forward without bending their knees. The new distance between the two points is measured again, 15 cm is subtracted, and the result is recorded.
Modified Schober's Test | 2 weeks
  It is a commonly used method for assessing lumbar mobility. The patient stands with their feet shoulder-width apart, and a mark is placed between two PSIS, adding 15 cm to it. The patient is then instructed to bend forward without bending their knees. The new distance between the two points is measured again, 15 cm is subtracted, and the result is recorded.
lumbar flexion range of motion | Baseline
  TiltMeter© app with an iPhone© could efficiently measure lumbar spine flexion ROM. The iPhone© is placed at T12-L1 and then at S1-S2 during maximum flexion of the lumbar spine. Total ROM is calculated by subtracting the S1-S2 measurement from T12-L1.
lumbar flexion range of motion | 30 minutes
  TiltMeter© app with an iPhone© could efficiently measure lumbar spine flexion ROM. The iPhone© is placed at T12-L1 and then at S1-S2 during maximum flexion of the lumbar spine. Total ROM is calculated by subtracting the S1-S2 measurement from T12-L1.
lumbar flexion range of motion | 2 weeks
  TiltMeter© app with an iPhone© could efficiently measure lumbar spine flexion ROM. The iPhone© is placed at T12-L1 and then at S1-S2 during maximum flexion of the lumbar spine. Total ROM is calculated by subtracting the S1-S2 measurement from T12-L1.
lumbar extension range of motion | Baseline
  TiltMeter© app with an iPhone© could efficiently measure lumbar spine extension ROM. The iPhone© is placed at T12-L1 and then at S1-S2 during maximum extension of the lumbar spine. Total ROM is calculated by subtracting the S1-S2 measurement from T12-L1.
lumbar extension range of motion | 30 minutes
  TiltMeter© app with an iPhone© could efficiently measure lumbar spine extension ROM. The iPhone© is placed at T12-L1 and then at S1-S2 during maximum extension of the lumbar spine. Total ROM is calculated by subtracting the S1-S2 measurement from T12-L1.
lumbar extension range of motion | 2 weeks
  TiltMeter© app with an iPhone© could efficiently measure lumbar spine extension ROM. The iPhone© is placed at T12-L1 and then at S1-S2 during maximum extension of the lumbar spine. Total ROM is calculated by subtracting the S1-S2 measurement from T12-L1.
Oswestry Low Back Pain Scale | Baseline
  The Oswestry Disability Index assesses various aspects of daily life functioning through 10 different categories, such as pain intensity, personal care, mobility, and social activities. Each category consists of 6 questions, with each question scored on a scale of 0 to 5. The total score ranges from 0 to 50, which can then be converted to a scale of 0 to 100.Higher values represent a worse outcome.
Oswestry Low Back Pain Scale | 30 minutes
  The Oswestry Disability Index assesses various aspects of daily life functioning through 10 different categories, such as pain intensity, personal care, mobility, and social activities. Each category consists of 6 questions, with each question scored on a scale of 0 to 5. The total score ranges from 0 to 50, which can then be converted to a scale of 0 to 100.Higher values represent a worse outcome.
Oswestry Low Back Pain Scale | 2 weeks
  The Oswestry Disability Index assesses various aspects of daily life functioning through 10 different categories, such as pain intensity, personal care, mobility, and social activities. Each category consists of 6 questions, with each question scored on a scale of 0 to 5. The total score ranges from 0 to 50, which can then be converted to a scale of 0 to 100.Higher values represent a worse outcome.
SF-36 | Baseline
  The scale evaluates quality of life across eight different subcategories: physical functioning, physical role difficulty, emotional role difficulty, energy, mental health, social functioning, pain, and general health perception. Each subcategory is scored between 0 and 100, Higher values represent a worse outcome.
SF-36 | 30 minutes
  The scale evaluates quality of life across eight different subcategories: physical functioning, physical role difficulty, emotional role difficulty, energy, mental health, social functioning, pain, and general health perception. Each subcategory is scored between 0 and 100, Higher values represent a worse outcome.
SF-36 | 2 weeks
  The scale evaluates quality of life across eight different subcategories: physical functioning, physical role difficulty, emotional role difficulty, energy, mental health, social functioning, pain, and general health perception. Each subcategory is scored between 0 and 100, Higher values represent a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University Institute of Health Sciences, Kartal, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
We have not decided yet, but at this moment, we decided to share brief data with future researchers after requesting and submitting ethical committee permission.

REFERENCES:
- [Background] Fernandes WVB, Blanco CR, Politti F, de Cordoba Lanza F, Lucareli PRG, Correa JCF. The effect of a six-week osteopathic visceral manipulation in patients with non-specific chronic low back pain and functional constipation: study protocol for a randomized controlled trial. Trials. 2018 Mar 2;19(1):151. doi: 10.1186/s13063-018-2532-8. PMID 29499728
- [Background] Santos GK, Goncalves de Oliveira R, Campos de Oliveira L, Ferreira C de Oliveira C, Andraus RA, Ngomo S, Fusco A, Cortis C, DA Silva RA. Effectiveness of muscle energy technique in patients with nonspecific low back pain: a systematic review with meta-analysis. Eur J Phys Rehabil Med. 2022 Dec;58(6):827-837. doi: 10.23736/S1973-9087.22.07424-X. Epub 2022 Sep 28. PMID 36169931
- [Background] Maharty DC, Hines SC, Brown RB. Chronic Low Back Pain in Adults: Evaluation and Management. Am Fam Physician. 2024 Mar;109(3):233-244. PMID 38574213
- [Background] Chun SW, Lim CY, Kim K, Hwang J, Chung SG. The relationships between low back pain and lumbar lordosis: a systematic review and meta-analysis. Spine J. 2017 Aug;17(8):1180-1191. doi: 10.1016/j.spinee.2017.04.034. Epub 2017 May 2. PMID 28476690
- [Background] Airaksinen O, Brox JI, Cedraschi C, Hildebrandt J, Klaber-Moffett J, Kovacs F, Mannion AF, Reis S, Staal JB, Ursin H, Zanoli G; COST B13 Working Group on Guidelines for Chronic Low Back Pain. Chapter 4. European guidelines for the management of chronic nonspecific low back pain. Eur Spine J. 2006 Mar;15 Suppl 2(Suppl 2):S192-300. doi: 10.1007/s00586-006-1072-1. No abstract available. PMID 16550448
- [Background] Park MW, Park SJ, Chung SG. Relationships Between Skeletal Muscle Mass, Lumbar Lordosis, and Chronic Low Back Pain in the Elderly. Neurospine. 2023 Sep;20(3):959-968. doi: 10.14245/ns.2346494.247. Epub 2023 Sep 30. PMID 37798990
- [Background] Jorgensson A. The iliopsoas muscle and the lumbar spine. Aust J Physiother. 1993;39(2):125-32. doi: 10.1016/S0004-9514(14)60477-3. PMID 25026138
- [Background] Lakkadsha TM, Qureshi MI, Kovela RK, Saifee SS, Lalwani SS. Efficacy of Single Stretching Session of Iliopsoas Using Proprioceptive Neuromuscular Facilitation Versus Muscle Energy Technique on Low Back Pain in Patients With Lumbar Hyper-Lordosis. Cureus. 2022 Aug 12;14(8):e27916. doi: 10.7759/cureus.27916. eCollection 2022 Aug. PMID 36110466
- [Background] Lifshitz L, Bar Sela S, Gal N, Martin R, Fleitman Klar M. Iliopsoas the Hidden Muscle: Anatomy, Diagnosis, and Treatment. Curr Sports Med Rep. 2020 Jun;19(6):235-243. doi: 10.1249/JSR.0000000000000723. PMID 32516195
- [Background] Siglan U, Colak S. Effects of diaphragmatic and iliopsoas myofascial release in patients with chronic low back pain: A randomized controlled study. J Bodyw Mov Ther. 2023 Jan;33:120-127. doi: 10.1016/j.jbmt.2022.09.029. Epub 2022 Sep 29. PMID 36775506
- [Background] Tanigawa MC. Comparison of the hold-relax procedure and passive mobilization on increasing muscle length. Phys Ther. 1972 Jul;52(7):725-35. doi: 10.1093/ptj/52.7.725. No abstract available. PMID 5034102
- [Background] Ashrafi A, Arab AM, Abdi S, Nourbakhsh MR. The association between myofascial trigger points and the incidence of chronic functional constipation. J Bodyw Mov Ther. 2021 Apr;26:201-206. doi: 10.1016/j.jbmt.2020.12.004. Epub 2020 Dec 3. PMID 33992245
- [Background] Wong CK. Strain counterstrain: current concepts and clinical evidence. Man Ther. 2012 Feb;17(1):2-8. doi: 10.1016/j.math.2011.10.001. Epub 2011 Oct 24. PMID 22030379
- [Background] Patel VD, Eapen C, Ceepee Z, Kamath R. Effect of muscle energy technique with and without strain-counterstrain technique in acute low back pain - A randomized clinical trial. Hong Kong Physiother J. 2018 Jun;38(1):41-51. doi: 10.1142/S1013702518500051. Epub 2018 Apr 4. PMID 30930578